CLINICAL TRIAL: NCT00091481
Title: A Randomized, Active-Controlled, Double-Blind Multi-Center Study to Compare Initial Dosing Parameters of Zemplar in Stage V Chronic Kidney Disease Subjects on Hemodialysis
Brief Title: Study to Compare Initial Dosing Parameters of Zemplar in Stage V Chronic Kidney Disease Subjects on Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01-367
Record Dates: First submitted 2004-09-09; First posted 2004-09-13 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Kidney Failure, Chronic
Keywords: Stage V Chronic Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — paricalcitol

INTERVENTIONS:
Drug: Zemplar

SUMMARY:
To show non-inferiority in the incidence rates of elevated calcium-phosphorus product between two treatment groups: 1) a group having an initial dose based on baseline PTH (baseline iPTH/80) and 2) a group having a starting dose based on body weight (0.04 mcg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Stage V Chronic Kidney Disease
* Patients on Hemodialysis requiring treatment for secondary hyperparathyroidism with vitamin D therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2003-06

PRIMARY OUTCOMES:
Incidence rate of at least two consecutive calcium-phosphorus product levels greater than 65.

SECONDARY OUTCOMES:
Evaluate the number of days to achieve the first of 2 consecutive > or = 30% decreases from baseline in PTH
The incidence rate for hypercalcemia
The incidence rate for hyperphosphatemia

CONTACTS AND LOCATIONS:
Overall Officials: Jin Tian, M.D., Study Director — Abbott
Locations (19):
- Greece (19):
  - Errikos Dynan Hospital, Ambelokipi, Athens
  - General Hospital of Athens, "G.Gennimatas", Cholargós, Athens
  - General Hospital of Attica "Sismanoglio", Marousi, Athens
  - "Hygeia" Diagnosis and Therapy Center, Marousi, Athens
  - General Hospital of Melissia "Amalia Fleming", Melíssia, Athens
  - General Hospital of Voula Askilpieion, Voula, Athens
  - General Hospital of Heraklion, Voutes, Heraklion, Crete
  - General Hospital Thessaloniki "Papanikolaou", Eksochi, Thessaloniki
  - General Hospital of Veria, Papagou Area, Veria
  - Blue Cross Clinic, Athens
  - Evgenidio Clinic, Athens
  - Regional General Hospital of Athens "Korgialeneio-Benakeio", Athens
  - General University Hospital of Alexandroupolis, Dragana
  - Regional General Hospital of Ioannina "Hatzikosta", Ioannina
  - General University Hospital Ioannina, Ioannina
  - General Hospital of Nikea "Agios Panteleimon", Nikea, Piraeus 18454,
  - General Hospital of Thessaloniki "Ahepa", Thessaloniki
  - General Hospital of Thessaloniki "Hippokrateion", Thessaloniki
  - General Hospital of Thessaloniki "Papageorgiou", Thessaloniki